CLINICAL TRIAL: NCT02813369
Title: An Observational Post-Authorisation Safety Study (PASS) of MOVENTIG® (Naloxegol) Among Patients Aged 18 Years and Older Treated With Opioids Chronically
Brief Title: Naloxegol Health Outcome Post Authorisation Safety Study
Status: Terminated | Type: Observational
Why Stopped: Not feasible to reach the required number of patient cases by the defined end of data collection milestone (Q4 2022) knowing that the study completion was planned by the end of 2023
Sponsor: Kyowa Kirin Pharmaceutical Development Ltd (Industry)
Responsible Party: Sponsor
Organization: Kyowa Kirin Co., Ltd. (Industry)
Other Study IDs: D3820R00009
Record Dates: First submitted 2016-06-07; First posted 2016-06-27 (Estimated); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Opioid Induced Constipation
MeSH Terms: conditions — Opioid-Induced Constipation | interventions — naloxegol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- naloxegol: patients exposed to naloxegol
  Interventions: Drug: naloxegol
- non-PAMORA laxative: patient exposed to non-peripherally acting mu-opioid receptor antagonist (PAMORA) laxative
  Interventions: Drug: non-PAMORA laxative

INTERVENTIONS:
Drug: naloxegol — non-interventional study where patients are exposed to naloxegol during normal clinical practice
  Groups: naloxegol
Drug: non-PAMORA laxative — non-interventional study where patients are exposed to non-peripherally acting mu-opioid receptor antagonist (PAMORA) laxative
  Groups: non-PAMORA laxative

SUMMARY:
This post-authorization observational safety study (PASS) monitors clinically important identified and potential risks within a cohort of patients treated with naloxegol, including the occurrence of bowel perforation, acute myocardial infarction (MI), stroke, cardiovascular (CV)-specific mortality, all-cause mortality, hypertension, opioid withdrawal, abdominal pain, diarrhea, syncope, and change in pain severity. This study is part of a broader post-marketing commitment to augment routine evaluation of the safety profile of naloxegol in clinical practice.

DETAILED DESCRIPTION:
The overall research goal for this study is to provide additional data to characterize the safety of naloxegol in the indicated population, grouped by cancer or non-cancer, and within at-risk vulnerable non-cancer populations identified in the naloxegol risk management plan (RMP) by describing type and frequency of identified and potential risks (including bowel perforation, acute MI, stroke, CV-specific mortality, all-cause mortality, hypertension, opioid withdrawal, abdominal pain, diarrhea, syncope, and change in pain severity) in patients ≥18 years of age who were treated with opioids chronically and subsequently treated with naloxegol in routine post-authorization use.

The primary objective of the study is to assess the incidence risk of bowel perforation, acute MI, stroke, all-cause mortality, and hypertension in patients treated with naloxegol (Naloxegol Inception Cohort, (NIC)), grouped by cancer or non cancer, a Concurrent Reference Cohort (CRC) by cancer or non-cancer, and by pre-specified non-cancer sub-populations that include patients aged ≥65 years, pregnant patients, patients with prior CV, patients with prior renal or hepatic impairment, patients with concurrent methadone use, and patients with concurrent use of cytochrome P450 (CYP) 3A inhibitors/inducer or P-glycoprotein (Pgp) modulators.

An exploratory objective of the study is to assess the incidence risk of CV-specific mortality, opioid withdrawal, abdominal pain, diarrhea, syncope, and change in pain severity in patients treated with naloxegol (NIC) grouped by cancer and non cancer, a CRC grouped by cancer or non cancer, and by pre-specified non-cancer sub-populations that include patients aged ≥65 years, pregnant patients, patients with prior cardiovascular risk, patients with prior renal or hepatic impairment, patients with concurrent methadone use, and patients with concurrent use of CYP3A inhibitors/inducer or Pgp modulators.

ELIGIBILITY:
Inclusion Criteria:

1. Patient receives a new prescription for naloxegol or a non-PAMORA laxative. (Note: Only non-PAMORA laxatives that are approved/marketed in the European Union at the time naloxegol is authorized are permitted.)

Exclusion Criteria:

1. Patients <18 years of age on cohort entry date
2. Patients with <1 year of continuous data available prior to cohort entry date
3. Patients without exposure to current regular opioid use defined by >30 days of opioid exposure within the 180 days prior to and inclusive of the cohort entry date
4. Patients with evidence of a cancer indicator (diagnosis or treatment) prior to cohort entry date
5. Exposure to PAMORA laxatives, alvimopan, methylnaltrexone, or naloxone + opioid combination (including fixed-dose combinations) prior to cohort entry date

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in the targeted European countries who receive prescriptions for naloxegol will be identified for inclusion in the naloxegol inception cohort, while patients in these countries who receive a prescription for a non-PAMORA laxative will be identified for inclusion in the concurrent reference cohort. All patients in this study will be ≥18 years of age; have ≥1 year of continuous data available; have exposure to current, regular opioid use; and have no prior exposure to PAMORA laxatives alvimopan, methylnaltrexone, or naloxone + opioid combination (including fixed-dose combinations).
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2021-11 (Actual); Study Completion 2021-11 (Actual)

PRIMARY OUTCOMES:
Presence (yes/no) of bowel perforation | Can occur anytime through study completion, given no fixed follow-up timepoints, which can range from 1 day to 7 years
  Presence of a diagnostic or procedure code
Presence (yes/no) of acute MI | Can occur anytime through study completion, given no fixed follow-up timepoints, which can range from 1 day to 7 years
  Presence of a diagnostic code for acute MI, a diagnostic code for electrocardiogram supportive of MI or cardiac enzyme lab tests with positive results
Presence (yes/no) of stroke | Can occur anytime through study completion, given no fixed follow-up timepoints, which can range from 1 day to 7 years
  Presence of a diagnostic code for cerebral, cerebellar haemorrhage or infarction, cerebral embolism, stroke or cerebrovascular accident
Presence (yes/no) of all-cause mortality | Can occur anytime through study completion, given no fixed follow-up timepoints, which can range from 1 day to 7 years
  Record of death
Presence (yes/no) of hypertension | Can occur anytime through study completion, given no fixed follow-up timepoints, which can range from 1 day to 7 years
  Presence of a hypertension (HT) diagnostic code where no record of HT or treatment for HT was observed in the baseline, or a record of change in HT treatment type or dose from baseline was observed.

SECONDARY OUTCOMES:
Presence of (yes/no) CV-specific mortality | Can occur anytime through study completion, given no fixed follow-up timepoints, which can range from 1 day to 7 years
  Record of death that indicates the cause was a CV event
Presence of (yes/no) opioid withdrawal | Can occur anytime through study completion, given no fixed follow-up timepoints, which can range from 1 day to 7 years
  Presence of a diagnosis or symptom code
Presence of (yes/no) abdominal pain | Can occur anytime through study completion, given no fixed follow-up timepoints, which can range from 1 day to 7 years
  Presence of a diagnosis or symptom code
Presence of (yes/no) diarrhea | Can occur anytime through study completion, given no fixed follow-up timepoints, which can range from 1 day to 7 years
  Presence of a diagnosis or symptom code
Presence of (yes/no) syncope | Can occur anytime through study completion, given no fixed follow-up timepoints, which can range from 1 day to 7 years
  Presence of a diagnosis code
Presence of (yes/no) change in pain severity | Can occur anytime through study completion, given no fixed follow-up timepoints, which can range from 1 day to 7 years
  At least a doubling in opioid dose based on the morphine milligram equivalents (MME) from baseline

OTHER OUTCOMES:
Demographic characteristics | Can occur anytime through study completion, given no fixed follow-up timepoints, which can range from 1 day to 7 years
  Age (years), Gender (male, female, missing), Body mass index (kg/m2, as continuous variable and categorical), Smoking status (Current smoker, Past smoker, Never smoker,
  Unknown), Geographic indicator (e.g., England, Scotland, Northern Ireland, Wales)
Time characteristics | Can occur anytime through study completion, given no fixed follow-up timepoints, which can range from 1 day to 7 years
  Total duration of medical history (as continuous), Calendar year of index date (2015, 2016, 2017, 2018, 2019, 2020, 2021), Time (months) since launch of naloxegol (October 2015 in the UK, December 2014 for the Netherlands) at index date (as continuous variable and categorical)
Opioid-induced Constipation Characteristics: Prior constipation diagnosis | Can occur anytime through study completion, given no fixed follow-up timepoints, which can range from 1 day to 7 years
  Prior constipation diagnosis, within the previous five years or from start of patients' history if this period is less than 5 years (yes/no)
Opioid-induced Constipation Characteristics: Type of prior opioid use | Can occur anytime through study completion, given no fixed follow-up timepoints, which can range from 1 day to 7 years
  Type of prior opioid use prior to and excluding the index date : natural opium alkaloids , phenylpiperidine derivatives, diphenylpropylamine derivatives, benzomorphan derivatives, oripavine derivatives, morphinan derivatives, methadone, other opioids including opioids used in combination, drugs used in opioid dependence excluding lofexidine
Opioid-induced Constipation Characteristics: Amount of prior opioid use per day | Can occur anytime through study completion, given no fixed follow-up timepoints, which can range from 1 day to 7 years
  Amount (in mg converted to morphine milligram equivalent [MME] dose) of prior opioid use per day was determined using the last prescription within 180 days prior to and excluding index date.
Opioid-induced Constipation Characteristics: The amount of opioid exposure within 180 days | Can occur anytime through study completion, given no fixed follow-up timepoints, which can range from 1 day to 7 years
  The amount of opioid exposure within 180 days prior to and excluding index was categorised in four groups: at or below the median, above the median, dose = 0 and a separate category for missing.
Opioid-induced Constipation Characteristics: Type of laxative use | Can occur anytime through study completion, given no fixed follow-up timepoints, which can range from 1 day to 7 years
  Type of prior laxative use (prescribed prior to and excluding index): softeners and emollients, contact laxatives, bulk forming laxatives, osmotically acting laxatives, saline laxatives, and other drugs for constipation (e.g., lubiprostone, linaclotide, methylnaltrexone, prucalopride and enemas).
Opioid-induced Constipation Characteristics: Strength of laxative use | Can occur anytime through study completion, given no fixed follow-up timepoints, which can range from 1 day to 7 years
  The last prescription of any laxative prior to Naloxegol/non-PAMORA prescription (index date) and within 180 days of index date (exclusive) was used to determine the strength. For every laxative treatment in the database the prescribed strength and the number of patients on this strength are reported.
Opioid-induced Constipation Characteristics: Pre-existing conditions and comorbidities | Can occur anytime through study completion, given no fixed follow-up timepoints, which can range from 1 day to 7 years
  Comorbidities were identified through diagnosis codes during patient's baseline period (yes/no) Prior conditions : Cardiovascular, Pulmonary, Prior conditions, Neurologic, Gastrointestinal, Endocrine, Rheumatologic, Psychiatric, Renal Disease, Hepatic disease, Cancer, Pain conditions, Miscellaneous, Charlson Comorbidity index.
Evaluation of patients biochemical measurements at baseline | Can occur anytime through study completion, given no fixed follow-up timepoints, which can range from 1 day to 7 years
  Exposure to naloxegol (or the concurrent reference laxative) started on the index date. The exposure end date was calculated by an algorithm used to derive continuous exposure.
  We utilised quantity and number of tablets per day to calculate the days of supply for each prescription; this was combined with the refill sequence of successive prescriptions to calculate duration of continuous exposure, average daily dose and cumulative dose over the study period.
  Alanine aminotransferase: ≤35 U/L (females) or 40 U/L (males); >35 U/L (females) or 40 U/L (males); missing Serum creatinine: 0.7 to 1.3 mg/dL for men and 0.6 to 1.1 mg/dL for women; below those values; above those values; missing.
  Aspartate aminotransferase: ≤35 U/L; >35 U/L; missing Serum bilirubin: ≤1.9 mg/dL; >1.9 mg/dL; missing Tumour specific marker information (e.g., eGFR, JAK2, BRCA, Multiple Endocrine Neoplasia mutation)
Healthcare resource utilization during 12 month baseline period prior to index date | Can occur anytime through study completion, given no fixed follow-up timepoints, which can range from 1 day to 7 years
  Total number of hospitalisations (excluding A&E admission) Total number of specialist referrals (all specialities categorised as specialist/surgeon, GP, nurse, other health professionals, centre/team and other) Total number of lab tests Total number of outpatient physician visits (GP surgery visits) Total number of prescriptions (only prescriptions in primary care in THIN)
History of GI surgery | Can occur anytime through study completion, given no fixed follow-up timepoints, which can range from 1 day to 7 years
  Other variables of interest: Covariates included in the study are those determined to be potential risk factors for a given outcome of interest or predictors of exposure
Exposure | Exposure to naloxegol or the concurrent reference laxative started on the index date. The exposure end date was calculated by an algorithm used to derive continuous exposure
  Exposure to naloxegol or the concurrent reference laxative started on the index date. The exposure end date was calculated by an algorithm used to derive continuous exposure. The algorithm utilised quantity (naloxegol or concurrent reference laxative strength and number of tablets) and number of tablets per day (when available) to calculate the days of supply for each prescription; this was combined with the refill sequence of successive prescriptions to calculate duration of continuous exposure, average daily dose and cumulative dose over the study period.
Prior and Concomitant Medications at Baseline | Can occur anytime through study completion, given no fixed follow-up timepoints, which can range from 1 day to 7 years
  Prior and concomitant medications: prior was defined as any medications prescribed during patients' baseline period excluding the index date. Concomitant medications was defined as ongoing treatments at the initiation of naloxegol prescription. Prior medication and concomitant medication are not mutually exclusive groups. The drugs were classified in the following groups:
  Cardiovascular disease/risk factor-indicated medications Psychiatric-indicated medications Neurologic-indicated medications Musculoskeletal-indicated medications Alimentary Tract and Metabolism medications Genito Urinary System medications and Sex Hormones Blood and Blood Forming Organ medications Respiratory System medications Anti-infectives for Systemic Use Opioids Non-opioid analgesics CYP3A inducer - including subgroups of mild, moderate and strong inducers CYP3A inhibitor - including subgroups of mild, moderate and strong inhibitors Pgp modulator Methadone

CONTACTS AND LOCATIONS:
Locations (2):
- Research Site, Utrecht, Netherlands
- Research Site, Sutton, Surrey, United Kingdom